CLINICAL TRIAL: NCT05406973
Title: Comparison Between the SBK Microkeratome Versus Femtosecond Laser in Flap Creation During LASIK Surgery for Myopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Collaborators: Eyecare Center (Other)
Responsible Party: Principal Investigator, Mona Medhat, Ophthalmologist, Kasr El Aini Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kasr AlAini Hospital
Record Dates: First submitted 2017-09-13; First posted 2022-06-07 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Refractive Surgery
Keywords: LASIK, SBK, femtolaser, flap creation, myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moria SBK microkeratome (Other): Comparative non randomized Interventional clinical study between SBK microkeratome versus femtosecond laser in flap creation during LASIK surgery for myopia
  Interventions: Device: SBK microkeratome versus femtosecond laser in flap creation
- 200-kHz Femtosecond laser system (Other): Comparative non randomized Interventional clinical study between SBK microkeratome versus femtosecond laser in flap creation during LASIK surgery for myopia
  Interventions: Device: SBK microkeratome versus femtosecond laser in flap creation

INTERVENTIONS:
Device: SBK microkeratome versus femtosecond laser in flap creation — prospective comparative non randomized interventional clinical study

SUMMARY:
LASIK is the most commonly performed refractive surgery worldwide. It has been shown to be safe and effective procedure with predictable results over long term follow ups. With the advancement of technology, sub-Bowman keratomileusis allows thin flap of approximately 100 microns thickness thus preserving thicker stromal bed as compared to conventional LASIK. The femtosecond laser corneal flap has th advantage of producing a flap of uniform thickness, adjustable flap diameter, relatively few complications. The disadvantages of this procedure is the high cost of surgery, development of bubbles in the corneal layer and anterior chamber which may affect pupil trackingduring the procedure. Despite the emergence of femtosecond laser-assisted flap creation, mechanical microkeratomes remain the preferred choice in the majority of developing countries. Recent studies have shown that SBK corneal flap has the same advantages as femtosecond laser flap regarding flap uniformity, regularity, and accuracy with less suction time and cost, but with its specific complications as well.

DETAILED DESCRIPTION:
It is a prospective comparative non randomized interventional clinical study

Primary outcomes of this study include:

1. Comparison between the SBK microkeratome versus Femtosecond laser in flap creation during LASIK surgery for myopia using anterior segment OCT (AS-OCT) 1 month after surgery in each group of patients.
2. Measuring corneal flap diameter using (AS-OCT)

Secondary outcomes:

1. Measuring uncorrected and best corrected visual acuity after 1 day, 1 week, 1 month postoperative.
2. Recording any related complications in each group.

ELIGIBILITY:
Inclusion Criteria:

* Myopes (from -1 to -9), with astigmatism up to -4, normal corneal topography, central corneal thickness (CCT) more than 500 microns, and stable refraction for at least 12 months.

Exclusion Criteria:

* CCT less than 500 microns, any ocular pathologies, one eyed patients, history of systemic disease, intraoperative complications, and abnormal corneal topography.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
flap thickness accuracy | 1 month post operative
  comparison between the accuracy of the SBK microkeratome versus Femtosecond laser in flap creation during LASIK surgery for myopia, 1 month after surgery using anterior segment OCT

SECONDARY OUTCOMES:
Visual Acuity measurment | 1day, 1 week, 1 month after surgery
  measuring UCVA and BCVA

CONTACTS AND LOCATIONS:
Overall Officials: Yehia Salah El Din, MD, Principal Investigator — Professor of Ophthalmology, Kasr Al Aini
Locations (1):
- Eye Care Center, Maadi, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No